CLINICAL TRIAL: NCT01695668
Title: Treatment of Ocular Graft-versus-Host Disease (GVHD) With Topical Loteprednol
Brief Title: Treatment of Ocular Graft-versus-Host Disease (GVHD) With Topical Loteprednol Etabonate 0.5%
Acronym: Lotemax_BMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Shahzad Mian, Terry J. Bergstrom Professor for Resident Education, Associate Professor, Cornea and External Disease, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lotemax_00045815
Record Dates: First submitted 2012-09-25; First posted 2012-09-28 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Dry Eyes
Keywords: Graft versus Host Disease (GVHD); dry eyes; Bone marrow transplant (BMT); Restasis; Lotemax
MeSH Terms: conditions — Dry Eye Syndromes; Graft vs Host Disease | interventions — Loteprednol Etabonate; Cyclosporins; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotemax (Experimental): Loteprednol Etabonate 0.5%
  Interventions: Drug: Lotemax
- Restasis (Active Comparator): Cyclosporine
  Interventions: Drug: Restasis

INTERVENTIONS:
Drug: Lotemax — Ophthalmic corticosteroid. It decreases inflammation of the eye
  Other Names: Loteprednol
  Arms: Lotemax
Drug: Restasis — Restasis is an immunosuppressive agent. Cyclosporine may reduce inflammation in the eye.
  Other Names: cyclosporine
  Arms: Restasis

SUMMARY:
The purpose of this research is to:

1. Evaluate the safety and efficacy of a steroid eye drop (Lotemax) in patients who have been diagnosed with graft-versus-host disease (GVHD), which is a complication that may occur after bone marrow transplant where the newly transplanted material attacks the patient's body and may cause eye dryness.
2. Assess the safety and efficacy of Lotemax in decreasing the eye's reaction to the process in GVHD before the patient undergoes bone marrow transplant.
3. Compare how well Lotemax works in decreasing the process in GVHD with an immunosuppressive eye drop (Restasis), which has been commonly used in the treatment of this condition.

DETAILED DESCRIPTION:
Allogeneic bone marrow or peripheral stem cell transplantation result in Graft-versus-Host disease. Ocular symptoms may be the first presentation of GVHD and may be seen in the absence of systemic manifestations. GVHD is categorized into acute and chronic forms as defined by 100 days after the transplant. Acute GVHD is characterized by dermatitis, hepatitis, and enteritis. Chronic GVHD involves the skin, mouth, liver, gastrointestinal tract, lungs, and eyes. Ocular GVHD is a common cause of dry eye symptoms in patients who have undergone bone marrow transplant (BMT), and can be defined as ocular surface disease in the context of GVHD. Dry eyes develop in 76% of acute GVHD patients and between 62.5% and 81.8% of chronic GVHD patients. Current treatment for ocular GVHD includes topical cyclosporine 0.05% (Restasis, Allergan). Topical loteprednol etabonate 0.5% (Lotemax, Bausch and Lomb) has been shown to be safe and efficacious in treatment of inflammatory ocular disorders, but has not been prospectively studied in ocular GVHD.

2. Hypothesis: We anticipate that topical loteprednol etabonate 0.5% will be safe and efficacious in treatment of ocular GVHD patients, and would add to the armamentarium of therapeutics for this disease. Further, by following the natural progression of the disease prior to a patient's Bone Marrow Transplant (BMT), we may elucidate a new standard of care for these patients - one that involves referral to an ophthalmologist before ocular GVHD symptoms arise.

ELIGIBILITY:
Inclusion Criteria:

Scheduled for allogenic bone marrow transplant

Exclusion Criteria:

Allergic reaction to loteprednol or cyclosporine, previous allogenic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad Mian, MD, Principal Investigator — University of Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lotemax | Restasis
Started | 38 | 37
Completed | 23 | 20
Not Completed | 15 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotemax | Restasis | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.06 (13.68) | 51.21 (14.44) | 52.64 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Progression of Dry Eye Severity
Description: Dry eye is one of the major symptoms of ocular GVHD in bone-marrow transplant recipients, worsening of dry eye symptoms may be indicative of worsening ocular GVHD conditions.
Time Frame: 1 year
Measure: Number; unit: patients with increased dry eye severity
Arm/Group | Lotemax | Restasis
Number analyzed (Participants) | 38 | 37
patients with increased dry eye severity | 15 | 12

ADVERSE EVENTS:
Groups:
- Lotemax: Loteprednol Etabonate 0.5%
  Lotemax
- Restasis: Cyclosporine
  Restasis
Arm/Group | Lotemax | Restasis
Serious Adverse Events (participants affected / at risk) | 9/38 | 17/37
Other Adverse Events (participants affected / at risk) | 15/38 | 12/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotemax (N=38) | Restasis (N=37)
death (Blood and lymphatic system disorders) | 9 (9) | 17 (17)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lotemax (N=38) | Restasis (N=37)
severe Dry eye (Eye disorders) | 15 (15) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No